CLINICAL TRIAL: NCT02909062
Title: Beyond Performance Status: Electronic Activity Monitoring to Assess Functional Activity of Patients With Gastrointestinal Malignancy During Chemotherapy
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 16-493
Record Dates: First submitted 2016-09-19; First posted 2016-09-21 (Estimated); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Gastrointestinal Cancer
Keywords: Electronic Activity Monitoring (EAM); 16-493
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Electronic Activity Monitoring (EAM): This is a prospective, observational study. The study aims to examine the role of EAM as an objective, assessment of patient fitness in patients receiving chemotherapy for gastrointestinal malignancy. Physical activity level measured by EAM will be compared with standard measurement tools used by the oncology community to predict chemotherapy tolerability.
  Interventions: Device: Electronic Activity Monitoring (EAM); Behavioral: Daily Questionnaire

INTERVENTIONS:
Device: Electronic Activity Monitoring (EAM) — All registered patients will receive a wearable EAM device that will measure their physical activity. Patients will wear this device around their wrist for the designated period of assessment. The EAM device has the potential to measure active minutes, number of steps, distance walked and number of floors climbed. For the purpose of this study the EAM data captured will focus on daily step count.
Behavioral: Daily Questionnaire — Participants will be asked to complete this self-administered, paper-based questionnaire each day that they are expected to wear the EAM device. The questionnaire was designed specifically for the purpose of this study. It consists of 5 items that ask about the patient's perceived level of physical activity and fatigue in each 24 hour period that they have worn the EAM device. The daily questionnaires will be optional; however each participant will be encouraged to complete them.

SUMMARY:
Electronic activity monitoring (EAM) devices are wearable electronic devices that monitor functional activity and provide personal feedback on activity progression. This study aims to determine if EAM can provide an objective, assessment of patient functional activity. The study will also examine the change in functional activity experienced by patients during the first cycle of chemotherapy. Another objective of the study will be to see if baseline functional activity and the change in functional activity that occurs during the first cycle of chemotherapy can be used to predict patient tolerability of subsequent cycles of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of gastrointestinal malignancy.
* Age ≥ 18 years
* Planned to receive systemic chemotherapy, either adjuvant chemotherapy, or neoadjuvant chemotherapy, or any new line of chemotherapy in the setting of advanced disease. Subjects may enroll prior to chemotherapy or during the first cycle of treatment.

Exclusion Criteria:

* Restricted mobility defined as dependence or anytime use of a walker or wheelchair in the past three months.
* Refusing systemic chemotherapy.
* Concurrent radiotherapy with chemotherapy
* Have received at least one cycle of chemotherapy in the current chemotherapy regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MSK clinic
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2020-08-21 (Actual); Study Completion 2020-08-21 (Actual)

PRIMARY OUTCOMES:
EAM Max Step-count On-Chemotherapy - EAM Max Step-count Pre-Chemotherapy | 1 year
  change in physical activity between pre-chemotherapy and on-chemotherapy by counting the steps

CONTACTS AND LOCATIONS:
Overall Officials: Armin Shahrokni, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/